CLINICAL TRIAL: NCT00159809
Title: A Multi-Center, Flexible Dose Study With A Double-Blind, Randomized, Placebo-Controlled Phase Followed By An Open-Label Phase To Evaluate The Impact Of Treatment With Sildenafil Citrate On The Symptoms Of Depression And Quality Of Life (Qol) Of Male Patients With Erectile Dysfunction (ED)
Brief Title: Efficacy Study Measuring The Impact Of Treatment With Viagra On The Depressive Symptoms Of Men With Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481110
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Impotence; Depression
MeSH Terms: conditions — Erectile Dysfunction; Depression | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Viagra (Sildenafil citrate)

SUMMARY:
This study will measure the impact of treatment with Viagra on the depressive symptoms and quality of life in men with erectile dysfunction who have untreated depressive symptoms meeting the DSM-IV criteria for dysthymia or depression not otherwise specified (NOS), including minor depressive symptoms but excluding any form of psychotic disorder.

ELIGIBILITY:
Inclusion Criteria:

* Men above age of majority with ED (SHIM score less than 21)
* Beck Depression Inventory II score between 14 and 28

Exclusion Criteria:

* Subjects with symptoms of mania or major depressive disorders as demonstrated by the Mini International Neuropsychiatric Interview (MINI)
* Subjects who require treatment with antipsychotics, mood stabilizers, antidepressant agents or lithium (concomitant use of benzodiazepines is allowed) or who has required treatment with any of the above medication within the past 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2004-03; Study Completion 2004-08

PRIMARY OUTCOMES:
Describe the effect of treatment with sildenafil on the depressive symptoms in subjects with ED as measured by the BDI II at the end of the double-blind phase

SECONDARY OUTCOMES:
Measure QoL improvement; Describe treatment effect on social motivation & behavior; Describe relationship between depression severity and ED; Describe effectiveness of sildenafil; Describe correlation between the SEX FX and the IIEF; Validate the PREFA

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer